CLINICAL TRIAL: NCT06052085
Title: Investigation of the Efficiency of Pain Neuroscience Education in Patients With Chronic Pain After Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gursen, Doc. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22059
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: Cronic pain; Side effect; Pain neuroscience education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (Active Comparator): Pain Neuroscience Education; Four sessions of education will be applied. The neurophysiology of pain and the ability of the nervous system to modulate the experience of pain will be explained to the patient.
  Standard Physiotherapy Program; Soft tissue mobilization will be applied to the upper extremity twice a week for 6 weeks.
  Upper extremity exercises including breathing, warming, stretching and strengthening will be performed twice a week for 6 weeks.
  Interventions: Other: Pain Neuroscience Education; Other: Standard Physiotherapy Program
- Biomedical Pain Education (Active Comparator): Biomedical Pain Education; 4 sessions of education will be applied in 6 weeks. Pain will be explained to the patient from a biological point of view.
  Standard Physiotherapy Program; Soft tissue mobilization will be applied to the upper extremity twice a week for 6 weeks.
  Upper extremity exercises including breathing, warming, stretching and strengthening will be performed twice a week for 6 weeks.
  Interventions: Other: Biomedical Pain Education; Other: Standard Physiotherapy Program

INTERVENTIONS:
Other: Pain Neuroscience Education — Four sessions of Pain Neuroscience Education will be applied. The neurophysiology of pain and the ability of the nervous system to modulate the experience of pain will be explained to the patient.
  Arms: Pain Neuroscience Education
Other: Biomedical Pain Education — 4 sessions of Biomedical Pain Education will be applied in 6 weeks. Pain will be explained to the patient from a biological point of view.
  Arms: Biomedical Pain Education
Other: Standard Physiotherapy Program — Soft tissue mobilization will be applied to the upper extremity twice a week for 6 weeks. Upper extremity exercises including breathing, warming, stretching and strengthening will be performed twice a week for 6 weeks.

SUMMARY:
Breast cancer is the most common type of cancer among women worldwide. Various side effects are seen after the treatments (surgery, chemotherapy, radiotherapy, etc.). Fatigue and pain are the most common and persistent side effects of breast cancer treatments. Pain management in patients currently undergoing breast cancer surgery: It consists of medical treatment, physiotherapy program and psychosocial practices. Psychosocial practices include educational interventions. The most widely used is Biomedical Education. Biomedical Education explains pain to the patient from a biological point of view and may be insufficient in curing and preventing chronic pain. The increase in the knowledge of pain physiology has revealed the modern neuroscience-based Pain Neuroscience Education. Pain Neuroscience Education explains the neurophysiology of pain and the ability of the nervous system to modulate the experience of pain. When we look at the literature, it has been seen that the lack of studies in which my Pain Neuroscience Education was applied in chronic pain after breast cancer surgery and the results of existing studies were contradictory. The aim of this study to compare the effects of Pain Neuroscience Education applied together with a standard physiotherapy program on pain, somatode function, psychological function and quality of life in patients with chronic pain after breast cancer surgery in a randomized desing. The hypotheses of this study are as follows; H1(1): The effect of Pain Neuroscience Education and Biomedical Education applied in addition to standard physiotherapy on pain-related outcomes (pain severity and disability) is different in patients with chronic pain after breast cancer surgery.

H1(2): The effect of Pain Neuroscience Education and Biomedical Education applied in addition to standard physiotherapy on somatosensory function (pressure pain threshold and mechanical perception threshold) is different in patients with chronic pain after breast cancer surgery. H1(3) : The effect of Pain Neuroscience Education and Biomedical Education applied in addition to standard physiotherapy on psychological state (psychological symptoms (stress, anxiety and depression), pain-related catastrophe) in patients with chronic pain after breast cancer surgery is different. H1(4) : Pain Neuroscience Education and Biomedical Education applied in addition to standard physiotherapy have different effects on quality of life in patients with chronic pain after breast cancer surgery. The patients were over the age of 18, diagnosed with breast cancer, had at least three months after primary cancer treatments (surgery, chemotherapy, radiotherapy), had pain in the upper extremity and shoulder region for more than three months, and were evaluated on the Visual Analogue Scale in terms of pain intensity in the last week. Patients who indicate at least 40 points out of 100 (VAS) will be included. The Mini Mental Test will be applied to individuals over 65 years of age in terms of cooperation suitability and those with a score of 24 and above will be included in the study. Cases who met the inclusion criteria and accepted to participate in the study will be randomly assigned to 2 separate groups according to the online computer-based block randomization list. Pain Neuroscience Education and standard physiotherapy program (soft tissue mobilization + exercise) will be applied to the individuals in the 1st group, and Biomedical Education and standard physiotherapy program (soft tissue mobilization + exercise) will be applied to the individuals in the 2nd group. The working period is 6 weeks. Individuals in the 1st group will receive 4 sessions of Pain Neuroscience Training, and 4 sessions of Biomedical Pain Training will be applied to the individuals in the 2nd group. Standard physiotherapy will be applied to the cases in both groups for 6 weeks, 2 sessions per week. In the first session of the treatment, individuals in both groups will be informed about the treatment process. Individuals will be evaluated in terms of research and outcome measurements twice, at the beginning of the study and at the end of the 6th week, in line with the control frequencies used routinely in the clinic. The assessment will take approximately 45 minutes for each individual. At the beginning of the study, demographic and physical characteristics of individuals, medical and surgical background (cancer history, treatments, number of sessions and/or cures), drugs used (type and dosage), and lifestyle characteristics (alcohol and smoking and regular physical activity/exercise habits) ) related information will be saved. In the evaluation; Visual Analogue Scale, Pain Disability Index, Digital Pressure Algometer, Semmes Weinstein Monoflames, Pain Disaster Scale, Depression, Anxiety-Stress Scale-21(DASS-21), Functional Assessment of Cancer Treatment-Breast ( FACT-B+4) scale will be used.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Women diagnosed with breast cancer
* Patients who have passed at least 3 months after their primary treatment such as surgery, radiotherapy, chemotherapy
* Women who have pain in the upper extremity and shoulder region for more than three months and have achieved at least 40 points out of 100 on the Visual Analogue Scale (VAS) in the last week

Exclusion Criteria:

* Patients with chronic pain in the upper extremity/shoulder before the diagnosis of breast cancer,
* Patients who have previously undergone a pain education program,
* Those with metastases, bilateral or recurrent breast cancer,
* Lack of cooperation in assessment and/or treatment and illiteracy,
* Patients who did not consent to the study and did not have an informed consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity of the upper extremity | Change in pain intensity from baseline up to the end of the 6th week
  In our study, Visual Analog Scale(VAS) will be used to measure subjectively perceived pain. The Visual Analogue Scale (VAS) is a horizontal line of 0-10 cm denoting the absence of pain at one end and the most severe pain possible at the other. The subjects will be asked to mark the pain they have experienced in the last 3 days on the VAS.
Pain Related Dysfunction | Change in pain-related dysfunction from baseline to end of week 6
  Pain Disability Questionnaire (PDQ) will be used to measure pain-related disability. The Pain Disability Questionnaire (PDQ) is a seven-item scale aiming to determine the functional losses related to the musculoskeletal system suffered by the patient due to pain. From the patient, by giving 0 to 10 points to all questions; are asked to rate the impact on daily living activities, including family-home responsibilities, leisure activities, occupation, social activities, sexuality, and self-care.
  The total score ranges from 0 to 70. If the result is over 40 points, it means high disability.

SECONDARY OUTCOMES:
Somatosensory function: Pressure Pain Threshold | Change in pressure pain threshold from baseline to end of 6 weeks
  A Digital Pressure Algometer will be used to evaluate the pressure pain threshold. Pressure pain threshold is the amount of pressure at which pressure perception is first perceived as painful. It is applied until the participant states the point where the pressure is perceived as painful for the first time by saying 'stop'. The average of the two measurements is taken. The pressure pain threshold will be evaluated at the points in the pectoral muscle region, the lateral trunk side, and the upper trapezius muscle.
Somatosensory function: Mechanical Detection Threshold | Change in mechanical detection threshold from baseline up to the end of the 6th week
  Semmes Weinstein Monofilaments will be used. The mechanical sensing threshold and the mechanical pain threshold will be measured. The mechanical sensing threshold is the point at which the stimulus is first felt. The mechanical pain threshold is the point at which the stimulus is first felt painful. It will be applied to the inner side of the upper arm, the lateral trunk side and the quadriceps muscle.
Psychological Function: Pain Related Catastrophization | Change in Pain Related Catastrophization from baseline to end of week 6
  The Pain Catastrophizing Scale (PCS) will be used to measure pain-related catastrophication. This scale is a 14-item scale developed to examine catastrophic factors such as rumination, magnification, and weakness that are effective in the mechanism of pain.
  PCS scores range from 0 to 52 points. It is understood that the higher the score, the higher the catastrophization.
Psychological Function:Psychological Symptoms | Change in psychological symptoms from baseline to end of week 6
  Psychological Symptoms will be measured using the Depression Anxiety-Stress Scale-21(DASS-21). This scale measures the level of depression, anxiety and stress. It consists of 21 items and seven items in each subscale.
Life Quality | Change in life quality from baseline to end of week 6
  Functional Assesment of Cancer Treatment (FACT-B+4) Scale Coster et al. to evaluate the effects of arm morbidity on quality of life after breast cancer surgery. It consists of 42 items and 6 subscales: physical well-being, social/family well-being, emotional well-being, functional well-being, breast cancer and arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumeysa Konokman, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Groef A, Penen F, Dams L, Van der Gucht E, Nijs J, Meeus M. Best-Evidence Rehabilitation for Chronic Pain Part 2: Pain during and after Cancer Treatment. J Clin Med. 2019 Jul 5;8(7):979. doi: 10.3390/jcm8070979. PMID 31284377
- [Background] Ling CC, Lui LY, So WK. Do educational interventions improve cancer patients' quality of life and reduce pain intensity? Quantitative systematic review. J Adv Nurs. 2012 Mar;68(3):511-20. doi: 10.1111/j.1365-2648.2011.05841.x. Epub 2011 Oct 17. PMID 21999358
- [Background] Manfuku M, Nishigami T, Mibu A, Yamashita H, Imai R, Tanaka K, Kitagaki K, Hiroe K, Sumiyoshi K. Effect of perioperative pain neuroscience education in patients with post-mastectomy persistent pain: a retrospective, propensity score-matched study. Support Care Cancer. 2021 Sep;29(9):5351-5359. doi: 10.1007/s00520-021-06103-1. Epub 2021 Mar 6. PMID 33677717
- [Background] Von Korff M, Jensen MP, Karoly P. Assessing global pain severity by self-report in clinical and health services research. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3140-51. doi: 10.1097/00007632-200012150-00009. No abstract available. PMID 11124730
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Background] Cathcart S, Winefield AH, Rolan P, Lushington K. Reliability of temporal summation and diffuse noxious inhibitory control. Pain Res Manag. 2009 Nov-Dec;14(6):433-8. doi: 10.1155/2009/523098. PMID 20011713
- [Background] Mucke M, Cuhls H, Radbruch L, Baron R, Maier C, Tolle T, Treede RD, Rolke R. Quantitative sensory testing (QST). English version. Schmerz. 2021 Nov;35(Suppl 3):153-160. doi: 10.1007/s00482-015-0093-2. PMID 26826097
- [Background] Suren M, Okan I, Gokbakan AM, Kaya Z, Erkorkmaz U, Arici S, Karaman S, Kahveci M. Factors associated with the pain catastrophizing scale and validation in a sample of the Turkish population. Turk J Med Sci. 2014;44(1):104-8. doi: 10.3906/sag-1206-67. PMID 25558568
- [Background] Ugurlu M, Ugurlu GK, Erten S, Ulusoy Kaymak S, Caykoylu A. Reliability and Factorial Validity of the Turkish Version of the Pain Disability Index in Rheumatic Patients With Chronic Pain. Arch Rheumatol. 2016 Apr 26;31(3):265-271. doi: 10.5606/ArchRheumatol.2016.5750. eCollection 2016 Sep. PMID 29900947